CLINICAL TRIAL: NCT06020768
Title: The Effect of Different Bed-Head Angles on the Haemodynamic Parameters of Intensive Care Patients
Brief Title: The Effect of Different Bed-Head Angles on the Haemodynamic Parameters of Intensive Care Patients Lying in the Supine Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Dilek Yilmaz, PhD, Associate Professor, Uludag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-3/28
Record Dates: First submitted 2023-08-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Thyroidectomy; Colon Surgery; Cholecystectomy; Inguinal Hernia
Keywords: Intensive care units; haemodynamic parameters; central venous pressure; supine position; bed-head angle
MeSH Terms: conditions — Hernia, Inguinal; Deception

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the different bed-head angles in the supine position (Experimental): The researcher brought the patient to the supine position with the bed-head at 0 degree, and immediately (minute 0) made haemodynamic measurements: central venous pressure, systolic and diastolic blood pressure, heart rate, breathing rate and peripheral oxygen saturation. It was taken into account that this could change haemodynamic parameters, and immediately after a 10-minute period of rest, the same haemodynamic measurements were repeated. After this, the bed-head was adjusted to an angle of 20 degree, and the same procedure was repeated, with measurements after 0 and 10 minutes. The same procedure was followed with the bed-head raised to 30 degree and then to 45 degree. In positioning the patients' bed-heads to different angles, a spirit level and a protractor were used.
  Interventions: Other: the bed-head was raised to an angle of 0, 20, 30 and 45 degrees

INTERVENTIONS:
Other: the bed-head was raised to an angle of 0, 20, 30 and 45 degrees — With each patient in the supine position, the bed-head was raised to an angle of 0, 20, 30 and 45 degrees without a pillow, and the haemodynamic parameters of central venous pressure, systolic and diastolic blood pressure, heart rate, breathing rate and peripheral oxygen saturation were recorded after 0 and 10 minutes.
  Other Names: haemodynamic parameters were recorded

SUMMARY:
Aim: The aim of this study was to examine the effect of different bed-head angles given to patients lying in the supine position in an intensive care unit on the haemodynamic parameters of central venous pressure, systolic and diastolic blood pressure, heart rate, breathing rate and peripheral oxygen saturation.

Methods: The study was conducted with 50 intensive care patients aged 18 and over in a general surgery intensive care unit in Turkey. With each patient in the supine position, the bed-head was raised to an angle of 0, 20, 30 and 45 degrees without a pillow, and the haemodynamic parameters of central venous pressure, systolic and diastolic blood pressure, heart rate, breathing rate and peripheral oxygen saturation were recorded after 0 and 10 minutes.

DETAILED DESCRIPTION:
Aim: The aim of this study was to examine the effect of different bed-head angles given to patients lying in the supine position in an intensive care unit on the haemodynamic parameters of central venous pressure, systolic and diastolic blood pressure, heart rate, breathing rate and peripheral oxygen saturation.

Design: This was a non-randomised quasi-experimental repeated measures study. Settings: The study was conducted with 50 intensive care patients aged 18 and over in a general surgery intensive care unit in Turkey.

Methods: With each patient in the supine position, the bed-head was raised to an angle of 0, 20, 30 and 45 degrees without a pillow, and the haemodynamic parameters of central venous pressure, systolic and diastolic blood pressure, heart rate, breathing rate and peripheral oxygen saturation were recorded after 0 and 10 minutes. The data obtained was evaluated using the Mann-Whitney test, the Kruskal Wallis test and the Bonferroni test.

ELIGIBILITY:
Inclusion Criteria:

* participating voluntarily in the study
* being aged over 18 years,
* having stayed in the General Surgery Intensive Care Unit for at least 24 hours,
* being monitored for 24 hours,
* having a central venous catheter inserted,
* having central venous pressure measured.

Exclusion Criteria:

* being less than 18 years of age,
* not wanting to participate in the study, or during the course of the research, wishing to withdraw from the study,
* receiving sedation treatment,
* receiving haemodialysis treatment,
* having an oxygen saturation value of less than 90%,
* being unable to tolerate a 0° prone position (hypovolemic or bradycardic).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
central venous pressure | 4 months
  central venous pressure in mmHg
blood pressure | 4 months
  blood pressure pressure in mmHg
heart rate | 4 months
  heart rate in beats
breathing rate | 4 months
  breathing rate in breaths
peripheral oxygen saturation | 4 months
  peripheral oxygen saturation in %

SECONDARY OUTCOMES:
weight | 4 months
  weight in kilograms
height | 4 months
  height in meters
BMI | 4 months
  BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University Hospital, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided